CLINICAL TRIAL: NCT06010927
Title: Ketamine/Midazolam Premedication Versus Pre-extubation Ketofol. Effect on Emergence Agitation and Recovery Profile After Pediatric Adenotonsillectomy: A Randomized Comparative Study.
Brief Title: Effect of Ketamine/Midazolam Premedication Versus Pre-extubation Ketofol on Recovery Profile in Pediatrics Undergoing Adenotonsillectomy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abeer Ahmed, MD, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-92-2023
Record Dates: First submitted 2023-06-28; First posted 2023-08-25 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Ketamine; Midazolam

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-A; ketamine/midazolam premedication (Active Comparator)
  Interventions: Drug: ketamine/midazolam
- Group-B: Ketofol pre-extubation (Active Comparator)
  Interventions: Drug: Ketofol

INTERVENTIONS:
Drug: ketamine/midazolam — premedication
  Arms: Group-A; ketamine/midazolam premedication
Drug: Ketofol — Pre-extubation
  Arms: Group-B: Ketofol pre-extubation

SUMMARY:
An optimum recovery profile after AT includes a rapid, smooth awakening without emergence agitation (EA), stable vital signs and oxygenation, reduced postoperative nausea and vomiting (PONV), controlled postoperative pain, and patient or parents' satisfaction. Ketamine is a low-cost drug with a wide therapeutic window. Ketamine is a competitive N-methyl-D-aspartate receptor antagonist with good analgesic properties and periprocedural amnesia.

The ketamine/midazolam combination was administered in different ways with controversial results about their effect on the EA and recovery profile.

Ketofol, a mixture of ketamine and propofol, has been used in different favorable recovery profiles regarding postoperative EA and PONV.

This study aims to evaluate the effect of premedication with an intramuscular ketamine/ midazolam combination versus pre-extubation ketofol on the EA and the recovery profile.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Children scheduled for AT under general anesthesia (GA).

Exclusion Criteria:

* Congenital cardiovascular anomalies
* Behavioral changes
* Delayed physical development
* Children receiving sedatives or anticonvulsants therapy

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
incidence of Emergence agitation | starting from time of PACU admission after recover from anesthesia till 6 hours postoperative

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Abeer Ahmed, Maadi, Cairo Governorate
  - Anesthesia department - Faculty of medicine- Cairo University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided